CLINICAL TRIAL: NCT04675229
Title: Extending the Validation and Reliability Testing of SCREEN: A Nutrition Risk Screening Tool for Community-living Seniors
Brief Title: Extending the Validation of SCREEN to Persons Living With Dementia or in Retirement Homes
Acronym: SCREEN
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Waterloo (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Heather Keller, Professor, University of Waterloo
Other Study IDs: ORE#42827
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-12

CONDITIONS: Malnutrition; Nutrition Poor; Dementia
Keywords: nutrition risk; dementia; retirement; validity; reliability
MeSH Terms: conditions — Malnutrition; Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Older adults (≥ 55 years) who do not eat enough nutritious food are at risk of malnutrition. Malnutrition can lead to frailty, hospitalization, poor quality of life, and death. SCREEN (Seniors in the Community Risk Evaluation for Eating and Nutrition) is the leading nutrition risk screening tool for cognitively well older adults living in the community. The purpose of this study is to determine if SCREEN can be used to find nutrition risk among older adults diagnosed with mild cognitive impairment or dementia (i.e., MCI-D) or those with a MoCA < 26 living in the community and persons living in retirement homes.

SCREEN and other nutrition and health measures will be completed in 600 older adults (300 living in retirement homes with or without MCI-D, and 300 living with MCI-D in the community). SCREEN will be completed twice to determine reliability, and persons with MCI-D will have their results compared to those of a caregiver who completes it on their behalf. A dietitian's assessment and rating of nutrition risk will be used as the gold-standard to determine validity.

DETAILED DESCRIPTION:
About a third of cognitively well, community-living older Canadians are at nutrition risk, which has been shown to lead to hospitalizations, poor quality of life, and death. Since SCREEN was created 20 years ago, there has been considerable growth in the number of community-living older adults diagnosed with mild cognitive impairment or dementia (i.e., MCI-D) and/or living in retirement homes. These two groups are nutritionally vulnerable. Nutrition risk is specifically associated with the progression of cognitive impairment and frailty, as well as caregiver burden. Yet, these groups are under-served with respect to nutrition care; dietitian services are not available in retirement homes and limited in many primary or memory care clinics. Nutrition screening and subsequent management of identified nutrition problems by accessing diverse community services (e.g., meal programs) in Canadian older adults is recommended because it can promote independence and delay frailty. However, preventative management for those with MCI-D or living in retirement homes is limited by lack of systematic nutrition screening with a valid and reliable tool that is feasible for these vulnerable seniors.

SCREEN is the leading nutrition risk tool for community-living seniors and is the logical choice for use in those with MCI-D and/or living in retirement residences. However, it has not been validated in these groups. It cannot be assumed that the existing validation in cognitively well older adults living in their own homes can translate to these two vulnerable groups. As well, one question on grocery shopping needs to be changed to accommodate persons living in retirement homes. This study is also timely with the recent update of Canada's Food Guide and recommendations to increase protein intake to mitigate frailty. Two questions on SCREEN need to be modified to adapt the new language on protein foods used in the new Food Guide. This study will undertake the validation and reliability testing of SCREEN, considering these minor revisions, in 600 older adults (community-dwelling older adults with MCI-D and those living in retirement homes with or without MCI-D). Validation of SCREEN for these populations will ensure that a single tool can be used in all older adults living in community and retirement settings. Specifically, understanding at what point a person with MCI-D is no longer a reliable informant for completing SCREEN will help with identification when a caregiver should complete the questionnaire. This is why the Montreal Cognitive Assessment is used, as it provides discrete scores differentiating mild cognitive impairment from dementia. The results of this study will have significant impact on practice by allowing, for the first time, confidence in the identification of nutrition risk in these under-served groups in Canada. There is an urgent need for this research. Early identification of nutrition risk and its subsequent management has the potential to advance our health care system by promoting the prevention of frailty and its consequences. This study will have a meaningful impact in the 'real world' setting of primary and community care for older adults in Canada and worldwide, by providing a feasible, validated and useful nutrition risk tool.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* potential participants with MCI-D will have a caregiver who either lives with the participant or is in daily contact OR
* potential participants have subjective complaint - MoCA used to confirm cogntive change OR
* Retirement home participants will have lived in their residence for a minimum of 3 months
* read and communicate in English
* provide written consent or assent for persons MCI-D; caregiver written consent required if participant with cognitive change unable to provide

Exclusion Criteria:

* living in a nursing home
* do not speak or read English
* live outside of the geographic boundaries of this study (i.e., > 45 km from Kitchener/Waterloo or London).

Min Age: 55 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Persons living with diagnosed dementia Persons with subjective complaint for memory and MoCA < 26 Persons living in a retirement home
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-09-25 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Validity of SCREEN | 3 years
  Comparison of SCREEN to a dietitian's assessment
Reliability of SCREEN | 3 years
  Test-retest reliability

CONTACTS AND LOCATIONS:
Overall Officials: Heather Keller, Principal Investigator — U Waterloo
Locations (1):
- Heather Keller, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Repository at University of Waterloo
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 2025- 2035
Access Criteria: University research